CLINICAL TRIAL: NCT00873860
Title: A Phase 2a, Randomized, Double-blind, Placebo-Controlled, Parallel-Arm, Multicenter Study to Evaluate the Efficacy and Safety of CAT-354, a Recombinant Human Monoclonal Antibody Directed Against Interleukin-13 (IL-13), on Asthma Control in Adults With Uncontrolled, Moderate-to-severe, Persistent Asthma
Brief Title: Study to Evaluate the Safety and Efficacy of CAT-354
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MI-CP199; 2008-007844-33 (EudraCT Number)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: CAT-354; Tralokinumab; Asthma
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo matched to CAT-354 subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Interventions: Other: Placebo
- CAT-354 150 mg (Experimental): CAT-354 150 milligram (mg) subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Interventions: Biological: CAT-354 150 mg
- CAT-354 300 mg (Experimental): CAT-354 300 mg subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Interventions: Biological: CAT-354 300 mg
- CAT-354 600 mg (Experimental): CAT-354 600 mg subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Interventions: Biological: CAT-354 600 mg

INTERVENTIONS:
Other: Placebo — Placebo matched to CAT-354 subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Arms: Placebo
Biological: CAT-354 150 mg — CAT-354 150 milligram (mg) subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Other Names: Tralokinumab
  Arms: CAT-354 150 mg
Biological: CAT-354 300 mg — CAT-354 300 mg subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Other Names: Tralokinumab
  Arms: CAT-354 300 mg
Biological: CAT-354 600 mg — CAT-354 600 mg subcutaneous injection once every 2 weeks on Day 1, 15, 29, 43, 57, 71, and 85.
  Other Names: Tralokinumab
  Arms: CAT-354 600 mg

SUMMARY:
This is a Phase 2a, randomized, double-blind, placebo-controlled, parallel-arm study to evaluate the efficacy and safety of 3 subcutaneous (SC) treatment regimens of CAT-354 in adult subjects with uncontrolled, moderate-to-severe, persistent asthma.

DETAILED DESCRIPTION:
Study MI-CP199, a Phase 2a, randomized, double-blind, placebo-controlled, parallel-arm, multicenter study will evaluate the effect of 3 SC treatment regimens of CAT-354 on asthma control in adults with uncontrolled, moderate-to-severe, persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Age 18 to 65 years at the time of Screening
* Subjects must have a body mass index (BMI) between 18 and 40 kilogram per square meter (kg/m^2)
* Written informed consent obtained from the subject prior to performing any protocol related procedures, including Screening evaluations
* Physician-diagnosed moderate-to-severe, persistent asthma requiring treatment with appropriate asthma controller medication
* Shows forced expiratory volume in 1 second (FEV1) reversibility postbronchodilator of greater than or equal to (>=)12 percent and >=200 milliliter (mL) or have shown such values in a previous test within the last year, or have a positive airway hyperresponsiveness (AHR) test result in the last year
* Pre-bronchodilator FEV 1 value >=40 percent of individual predicted value at Visits 1 and 3
* Uncontrolled asthma consistent with Expert Panel Report (EPR)-3. In the 2 to 4 weeks preceding Screening, subjects should have a history of 1 or more of the following: Daytime asthma symptoms >=2 days/week, Nighttime awakening >=1 night/week, Salbutamol use >=2 days/week
* An Asthma control questionnaire (ACQ) score >=1.5 at Visits 1 and 3
* At least 1 occurrence of asthma exacerbation in the past year that required an unscheduled medical encounter
* Men, unless surgically sterile, must likewise practice 2 effective methods of birth control (condom with spermicide) and must use such precautions from Day 1 through Study Day 169
* Otherwise healthy by medical history and physical examination for that age group
* A chest x-ray or computed tomography (CT) scan within the previous 12 months with no findings suggestive of acute or chronic respiratory pathology other than asthma
* Ability and willingness to complete the follow-up period until Day 169 as required by the protocol.

Exclusion Criteria:

* Known history of allergy or reaction to any component of the investigational product formulation
* Acute illness other than asthma at the start of the study
* History of an active infection within 4 weeks prior to Screening, or evidence of clinically significant active infection, including ongoing chronic infection
* History of ingestion of untreated water in a location known to be infected with parasites, resulting in acute or chronic diarrhea; or a diagnosis of parasitic infection within 6 months prior to Screening
* Use of immunosuppressive medication (except oral prednisone up to 10 milligram/day (mg/day) and inhaled and topical corticosteroids) within 30 days before randomization into the study
* Receipt of immunoglobulin or blood products within 30 days before randomization into the study
* Receipt of any investigational drug therapy or use of any biologicals including omalizumab within 6 months before the first dose of investigational product in this study or within 5 half-lives of an investigational agent or biologic, whichever is longer
* History of any known immunodeficiency disorder
* A positive hepatitis B surface antigen, or hepatitis C virus antibody
* A positive human immunodeficiency virus test or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report
* A live or attenuated vaccination received within 4 weeks prior to Screening
* Previous medical history, or evidence, of an intercurrent illness that may compromise the safety of the subject in the study
* History of clinically significant abnormality on electrocardiogram (ECG) in the opinion of the investigator
* Lactation (women)
* History of treatment for alcohol or drug abuse within the past year
* History suggestive of chronic obstructive pulmonary disease (COPD) and of cigarette smoking >=10 pack-years
* Evidence of any systemic disease on physical examination
* History of cancer, apart from basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy less than or equal to (<=)1 year prior to Study Day 1 or other malignancies treated with apparent success with curative therapy <=5 years prior to entry
* Known exposure to inhaled occupational agents or fumes
* Any condition (eg, cystic fibrosis [CF] or COPD) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of study results
* Individuals who are legally institutionalized
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or family members of such individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (34):
- Bulgaria (8):
  - Research Site, Burgas
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Sofia III
  - Research Site, Sofia II
  - Research Site, Stara Zagora
  - Research Site, Varna
- Germany (5):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Landsberg A. Lech
  - Research Site, Lich
  - Research Site, Mainz
- Poland (11):
  - Research Site, Bielsko-Biala
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Pikary Slaskie
  - Research Site, Skalskie
  - Research Site, Warsaw
  - Research Site, Warsazawa
  - Research Site, Warszawa II
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zabrze II
- Romania (6):
  - Research Site, Arad
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Deva
  - Research Site, Timisoara Timis
  - Research Site, Timișoara
- United Kingdom (4):
  - Research Site, Wythenshawe, Manchester
  - Research Site, Cambridge
  - Research Site, Leicester
  - Research Site, Manchester

REFERENCES:
- [Background] Piper E, Brightling C, Niven R, Oh C, Faggioni R, Poon K, She D, Kell C, May RD, Geba GP, Molfino NA. A phase II placebo-controlled study of tralokinumab in moderate-to-severe asthma. Eur Respir J. 2013 Feb;41(2):330-8. doi: 10.1183/09031936.00223411. Epub 2012 Jun 27. PMID 22743678
- [Derived] Baverel PG, White N, Vicini P, Karlsson MO, Agoram B. Dose-Exposure-Response Relationship of the Investigational Anti-Interleukin-13 Monoclonal Antibody Tralokinumab in Patients With Severe, Uncontrolled Asthma. Clin Pharmacol Ther. 2018 May;103(5):826-835. doi: 10.1002/cpt.803. Epub 2017 Sep 28. PMID 28758192
- [Derived] Wilkes DS, Chew T, Flaherty KR, Frye S, Gibson KF, Kaminski N, Klemsz MJ, Lange W, Noth I, Rothhaar K. Oral immunotherapy with type V collagen in idiopathic pulmonary fibrosis. Eur Respir J. 2015 May;45(5):1393-402. doi: 10.1183/09031936.00105314. Epub 2015 Jan 22. PMID 25614165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 357 participants were screened in this study, out of which 194 participants me the eligibility criteria and were enrolled and randomized into the study.
Period: Overall Study
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Started | 48 | 47 | 51 | 48
Treated | 47 | 47 | 51 | 48
Completed | 44 | 47 | 48 | 47
Not Completed | 4 | 0 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg | Total
Number analyzed (Participants) | 48 | 47 | 51 | 48 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.8) | 43.4 (11.1) | 48.7 (11.0) | 49.8 (10.4) | 47.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 19 | 36 | 28 | 116
  Male | 15 | 28 | 15 | 20 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Mean Asthma Control Questionnaire (ACQ) Score at Day 92
Description: Asthma Control Questionnaire (ACQ) is a participant-reported questionnaire to assess the asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Each item was rated on a 7-point Likert scale ranging from 0 (no impairment) to 6 (maximum impairment). Overall ACQ score is the mean of the 6 item scores with a score range of 0 (well controlled) to 6 (extremely poor controlled). Data collected on Day 1 prior to dosing was considered as baseline. Results were reported for overall ACQ score.
Time Frame: Day 1 and 92
Population: Evaluable population included all participants who received at least 4 doses of investigational product or received at least 1 dose but discontinued prior to receiving 4 doses due to safety reasons. Here, 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
units on a scale
  Day 1 (n=46, 46, 50, 47) | 2.63 (0.51) | 2.72 (0.58) | 2.62 (0.50) | 2.72 (0.76)
  Change at Day 92 (n= 46, 46, 51, 47) | -0.61 (0.90) | -0.73 (1.12) | -0.70 (0.93) | -0.86 (1.09)
Statistical Analysis 1: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 0.573, ANOVA — Change at Day 92: p-value was based on analysis of variance (ANOVA)
Statistical Analysis 2: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.640, ANOVA — Change at Day 92: p-value was based on ANOVA
Statistical Analysis 3: Comparison: Placebo vs CAT-354 600 mg; Test type: Superiority or Other; p = 0.224, ANOVA — Change at Day 92: p-value was based on ANOVA

2. Secondary Outcome: Time to First Observed Asthma Control
Description: Time to first asthma control was defined as the number of days from Study Day 1 to the post-baseline ACQ score measurement time point when greater than or equal to (>=) 0.5 reduction from baseline in mean ACQ score was first observed. Time to first asthma control was analyzed from Day 1 through Day 92 and up to entire study duration through Day 169. The ACQ score is a participant-reported questionnaire to assess the asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Each item was rated on a 7-point Likert scale ranging from 0 (no impairment) to 6 (maximum impairment). Overall ACQ score is the mean of the 6 item scores with a score range of 0 (well controlled) to 6 (extremely poor controlled).
Time Frame: Day 1 to Day 92 and Day 169
Population: Evaluable population = all participants who received at least 4 doses of investigational product or received at least 1 dose but discontinued treatment due to safety reasons. Since, >50% participants for each arm achieved improvement through Day 92; the median time-to-first observed achievement is identical for data through Day 92 and Day 169.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
days
  Day 1 to 92 | 25.5 (5.50) [15.0 to 71.0] | 22.0 (5.21) [15.0 to 43.0] | 15.0 (4.54) [15.0 to 43.0] | 15.0 (4.56) [15.0 to 36.0]
  Day 1 to 169 | 25.5 (9.97) [15.0 to 71.0] | 22.0 (8.89) [15.0 to 43.0] | 15.0 (7.65) [15.0 to 43.0] | 15.0 (8.07) [15.0 to 36.0]
Statistical Analysis 1: Comparison: Placebo vs CAT-354 150 mg; P-value were calculated with log-rank test, which was constructed by computing the observed and expected number of events (defined as achieving improvement from baseline in mean ACQ-6 score >= 0.5) at each observed event time and added to obtain an overall summary across all-time points where there was an event. Number of events was different for data through Day 92 comparing with data through Day 169. Therefore, the p-values were different for data through Day 92 and Day 169; Test type: Superiority or Other; p = 0.4686, Log Rank — Day 1 to 92: P-value was calculated against placebo group from a stratified log-rank test with atopic asthma status and tertile of baseline mean ACQ score as the stratification factors
Statistical Analysis 2: Comparison: Placebo vs CAT-354 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3170, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs CAT-354 600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1664, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs CAT-354 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3234, Log Rank — Day 1 to 169: P-value was calculated against placebo group from a stratified log-rank test with atopic asthma status and tertile of baseline mean ACQ score as the stratification factors
Statistical Analysis 5: Comparison: Placebo vs CAT-354 300 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3133, Log Rank — [p-value comment as in outcome 2, analysis 4]
Statistical Analysis 6: Comparison: Placebo vs CAT-354 600 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2108, Log Rank — [p-value comment as in outcome 2, analysis 4]

3. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Recorded at Study Sites at Day 1, 15, 29, 43, 57, 71, 85, 92, 127 and 169
Description: Forced Expiratory Volume in 1 Second (FEV1) is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Spirometry was performed with the participant in the sitting/standing (kept consistent at each visit) position at study sites by the investigator or qualified designee according to American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines. Multiple forced expiratory efforts (at least 3 but no more than 8) were performed for each office spirometry session and the 2 best efforts that met ATS/ERS acceptability and reproducibility criteria were recorded. The best efforts were based on the highest FEV1. The maximum FEV1 of the 2 best efforts was used for the analysis. Data collected on Day 1 prior to dosing was considered as baseline.
Time Frame: Day 1, 15, 29, 43, 57, 71, 85, 92, 127 and 169
Population: Evaluable population included all participants who received at least 4 doses of investigational product or received at least 1 dose but discontinued treatment due to safety reasons. Here, 'n' signifies those participants who were evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
liters
  Day 1 (n=46,46,51,47) | 1.949 (0.479) | 2.178 (0.661) | 1.907 (0.586) | 1.977 (0.646)
  Change at Day 15 (n=44,46,50,46) | 0.019 (0.420) | 0.122 (0.316) | 0.116 (0.378) | 0.134 (0.348)
  Change at Day 29 (n=46,46,49,47) | 0.051 (0.424) | 0.138 (0.315) | 0.149 (0.303) | 0.222 (0.354)
  Change at Day 43 (n=45,44,47,47) | 0.125 (0.399) | 0.131 (0.380) | 0.164 (0.358) | 0.147 (0.373)
  Change at Day 57 (n=45,46,49,47) | 0.043 (0.436) | 0.127 (0.339) | 0.187 (0.349) | 0.201 (0.344)
  Change at Day 71 (n=45,45,49,47) | 0.047 (0.397) | 0.158 (0.314) | 0.179 (0.381) | 0.190 (0.335)
  Change at Day 85 (n=45,46,48,47) | 0.087 (0.397) | 0.135 (0.342) | 0.286 (0.393) | 0.265 (0.473)
  Change at Day 92 (n=42,44,49,44) | 0.063 (0.476) | 0.158 (0.348) | 0.211 (0.374) | 0.262 (0.408)
  Change at Day 127 (n=44,44,49,47) | 0.094 (0.489) | 0.144 (0.263) | 0.241 (0.381) | 0.237 (0.285)
  Change at Day 169 (n=42,42,47,47) | 0.101 (0.442) | 0.204 (0.378) | 0.211 (0.394) | 0.236 (0.366)

4. Secondary Outcome: Change From Baseline in Peak Expiratory Flow (PEF) Recorded at Home Every Week From Day 1 to 169
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Home peak flow testing for PEF was performed every morning while sitting or standing prior to using any medication (if needed) for asthma. Mean of the data was collected over 1 week prior to dosing on Day 1 was considered as baseline. Mean PEF values for each week were used to calculate the change from baseline values starting from Day 2 to 169.
Time Frame: Day -7 to 1 (predose), Day 2 to 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
liters/minute
  Day -7 to 1 (n=46,46,51,47) | 282.63 (100.65) | 351.06 (130.41) | 291.54 (119.46) | 325.23 (123.90)
  Change in Day 2 to 8 (n=44,46,51,47) | -5.77 (22.74) | 1.91 (23.81) | -4.53 (19.02) | 5.94 (29.93)
  Change in Day 9 to 15 (n=45,46,51,47) | -7.46 (29.68) | -4.10 (28.15) | -2.83 (24.40) | 5.75 (42.34)
  Change in Day 16 to 22 (n=45,46,51,47) | -8.94 (35.72) | -6.53 (32.70) | -0.37 (33.85) | 10.55 (51.26)
  Change in Day 23 to 29 (n=44,46,51,47) | -10.53 (40.06) | -6.61 (37.95) | -0.79 (36.94) | 10.61 (52.64)
  Change in Day 30 to 36 (n=45,46,51,47) | -5.69 (44.69) | -5.69 (41.87) | -1.98 (36.06) | 6.52 (50.15)
  Change in Day 37 to 43 (n=44,46,50,47) | -11.08 (41.52) | -2.00 (49.76) | -4.07 (39.80) | 5.55 (54.28)
  Change in Day 44 to 50 (n=44,46,50,47) | -6.37 (41.50) | -9.02 (47.51) | -5.30 (36.57) | -0.84 (50.67)
  Change in Day 51 to 57 (n=45,46,50,47) | -7.00 (41.70) | -6.01 (47.36) | -4.85 (41.27) | -3.57 (52.84)
  Change in Day 58 to 64 (n=45,46,50,46) | -9.84 (38.73) | -2.83 (47.42) | -1.42 (41.90) | -0.73 (55.98)
  Change in Day 65 to 71 (n=45,46,50,46) | -11.81 (43.87) | -3.98 (47.20) | -0.92 (49.95) | -1.82 (49.79)
  Change in Day 72 to 78 (n=44,45,50,47) | -3.72 (44.07) | -3.42 (53.55) | 2.54 (45.58) | 1.78 (49.45)
  Change in Day 79 to 85 (n=45,45,50,46) | -10.83 (43.99) | -6.67 (54.49) | -0.35 (40.29) | 5.30 (60.62)
  Change in Day 86 to 92 (n=45,46,50,47) | -3.26 (47.36) | -6.66 (51.23) | 5.04 (40.52) | 0.31 (62.86)
  Change in Day 93 to 99 (n=45,46,50,47) | -2.52 (47.94) | -4.99 (49.91) | 5.16 (40.99) | 7.81 (58.29)
  Change in Day 100 to 106 (n=44,46,49,47) | -9.60 (55.47) | -7.33 (52.64) | 1.93 (43.08) | 2.00 (62.18)
  Change in Day 107 to 113 (n=44,45,48,47) | -7.53 (56.29) | -11.29 (57.33) | 0.53 (45.60) | 0.39 (61.52)
  Change in Day 114 to 120 (n=42,45,47,47) | -2.19 (61.74) | -8.97 (55.61) | 4.85 (39.54) | -3.03 (59.68)
  Change in Day 121 to 127 (n=42,46,46,46) | -3.58 (65.64) | -8.99 (64.60) | 3.61 (46.18) | -4.21 (57.88)
  Change in Day 128 to 134 (n=42,45,45,47) | -4.39 (61.22) | -14.81 (61.39) | 4.62 (44.65) | -2.64 (56.87)
  Change in Day 135 to 141 (n=40,45,47,47) | -0.26 (58.83) | -17.03 (58.99) | 1.11 (44.36) | -6.03 (63.13)
  Change in Day 142 to 148 (n=40,45,47,47) | 5.16 (66.54) | -11.63 (61.02) | -2.69 (51.65) | -9.65 (65.62)
  Change in Day 149 to 155 (n=40,45,46,47) | 0.43 (60.53) | -9.56 (60.13) | -7.65 (47.44) | -11.07 (62.16)
  Change in Day 156 to 162 (n=40,45,46,46) | -1.38 (65.53) | -11.60 (62.14) | -10.05 (43.11) | -10.68 (66.86)
  Change in Day 163 to 169 (n=37,41,42,40) | -0.36 (58.66) | -5.68 (60.69) | -4.71 (49.29) | -3.23 (66.84)

5. Secondary Outcome: Number of Puffs of Rescue Beta-2 Agonist Per Week
Description: Number of Puffs of Rescue Beta-2 Agonist Per Week Rescue beta-2 agonist use (total number of puffs for the preceding week) was collected daily in the morning by the participants in the daily diary provided to them. Average values for each week were reported starting from Day -7 to Day 169.
Time Frame: Day -7 to 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: puffs per week
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
puffs per week
  Day -7 to 1 (n=46,46, 51,47) | 2.58 (1.70) | 2.84 (2.03) | 2.04 (1.51) | 2.62 (1.96)
  Day 2 to 8 (n=45,46, 51,47) | 2.5 (1.8) | 2.4 (2.0) | 1.9 (1.5) | 2.3 (2.0)
  Day 9 to 15 (n=46,46, 51,47) | 2.4 (1.8) | 2.5 (2.3) | 1.9 (1.5) | 2.2 (2.0)
  Day 16 to 22 (n=46,46, 51,47) | 2.6 (1.9) | 2.2 (2.0) | 1.9 (1.7) | 2.3 (2.2)
  Day 23 to 29 (n=45,46, 51,47) | 2.7 (2.1) | 2.2 (2.0) | 2.0 (1.9) | 2.2 (2.1)
  Day 30 to 36 (n=46,46, 51,47) | 2.5 (2.0) | 2.1 (2.2) | 1.9 (2.0) | 2.0 (1.9)
  Day 37 to 43 (n=45,46, 50,47) | 2.4 (2.0) | 2.1 (2.2) | 1.9 (2.0) | 2.0 (2.0)
  Day 44 to 50 (n=45,46, 50,47) | 2.5 (2.0) | 1.9 (2.2) | 1.7 (2.0) | 2.0 (2.0)
  Day 51 to 57 (n=45,46, 50,47) | 2.5 (2.1) | 2.0 (2.0) | 1.8 (1.9) | 2.0 (2.1)
  Day 58 to 64 (n=46,46, 49,46) | 2.5 (2.2) | 1.9 (2.0) | 1.9 (2.0) | 1.8 (2.0)
  Day 65 to 71 (n=46,46, 50,47) | 2.7 (2.3) | 2.0 (2.0) | 1.8 (2.0) | 2.0 (1.9)
  Day 72 to 78 (n=45,45, 50,46) | 2.5 (2.2) | 2.0 (2.0) | 1.8 (2.1) | 1.9 (1.8)
  Day 79 to 85 (n=46,46, 50,46) | 2.6 (2.3) | 2.1 (2.1) | 1.9 (2.0) | 1.8 (1.8)
  Day 86 to 92 (n=46,46, 50,47) | 2.5 (2.3) | 2.0 (2.1) | 1.8 (2.0) | 1.7 (1.7)
  Day 93 to 99 (n=46,46, 50,47) | 2.4 (2.2) | 1.7 (2.0) | 1.8 (2.1) | 1.6 (1.8)
  Day 100 to 106 (n=45,46, 49,47) | 2.3 (2.1) | 1.9 (2.2) | 1.7 (2.2) | 1.8 (1.8)
  Day 107 to 113 (n=45,45, 48,47) | 2.4 (2.1) | 1.9 (2.2) | 1.7 (1.9) | 1.7 (1.6)
  Day 114 to 120 (n=43,45, 47,47) | 2.3 (2.0) | 1.9 (2.1) | 1.7 (1.9) | 1.7 (1.7)
  Day 121 to 127 (n=43,46, 46,47) | 2.2 (1.9) | 1.9 (2.2) | 1.8 (2.0) | 1.6 (1.6)
  Day 128 to 134 (n=44,45, 47,47) | 2.2 (2.1) | 1.8 (2.0) | 1.6 (1.9) | 1.6 (1.7)
  Day 135 to 141 (n=42,45, 47,47) | 2.2 (2.0) | 1.9 (1.9) | 1.7 (2.0) | 1.7 (1.8)
  Day 142 to 148 (n=42,45, 47,47) | 2.3 (2.0) | 1.9 (2.1) | 1.8 (2.0) | 1.8 (1.8)
  Day 149 to 155 (n=42,45, 46,47) | 2.4 (2.2) | 1.9 (2.1) | 1.8 (2.0) | 1.8 (1.8)
  Day 156 to 162 (n=42,45, 46,46) | 2.3 (2.1) | 1.9 (2.1) | 1.7 (2.2) | 2.0 (2.0)
  Day 163 to 169 (n=39,41,42,40) | 2.7 (2.6) | 1.9 (2.1) | 1.6 (1.8) | 1.7 (1.9)

6. Secondary Outcome: Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]) Scores
Description: Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]): a 32-item questionnaire that measures the functional impairments experienced by adult participants including 4 domains (Symptoms, Activity Limitations, Emotional Function, and Environmental Stimuli). Participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score was calculated as the mean response to all questions. The 4 domain scores were the means of the responses to the questions in each of the domains. Overall AQLQ score and 4 domain scores ranged from 7 (no impairment) to 1 (severe impairment).
Time Frame: Day 1, 29, 57, 92, 127 and 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
units on a scale
  Overall : Day 1 (n=41,41,44,39) | 4.22 (0.83) | 3.96 (0.89) | 4.12 (0.80) | 4.11 (0.94)
  Overall: Day 29 (n=43,41,44,40) | 4.39 (1.04) | 4.39 (1.01) | 4.47 (0.97) | 4.60 (0.91)
  Overall: Day 57 (n=44,40,43,45) | 4.57 (1.03) | 4.56 (1.15) | 4.47 (1.05) | 4.73 (0.96)
  Overall: Day 92 (n=40,42,40,38) | 4.70 (1.16) | 4.88 (1.31) | 4.74 (1.15) | 4.87 (0.99)
  Overall: Day 127 (n=41,42,44,42) | 4.69 (1.22) | 4.76 (1.29) | 4.64 (1.11) | 4.85 (1.13)
  Overall: Day 169 (n=41,44,45,44) | 4.72 (1.29) | 4.73 (1.26) | 4.61 (1.27) | 4.76 (1.13)
  Symptom: Day 1 (n=41,41,44,39) | 4.15 (0.88) | 3.89 (0.84) | 4.11 (0.71) | 4.08 (1.06)
  Symptom: Day 29 (n=43,41,44,40) | 4.32 (1.08) | 4.44 (1.07) | 4.48 (0.94) | 4.56 (1.01)
  Symptom: Day 57 (n=44,40,43,45) | 4.61 (1.02) | 4.68 (1.23) | 4.49 (1.05) | 4.73 (1.05)
  Symptom: Day 92 (n=40,42,40,38) | 4.77 (1.17) | 4.88 (1.40) | 4.78 (1.17) | 4.92 (1.01)
  Symptom: Day 127 (n=41,42,44,42) | 4.74 (1.33) | 4.79 (1.31) | 4.69 (1.09) | 4.95 (1.31)
  Symptom: Day 169 (n=41,44,45,44) | 4.82 (1.30) | 4.76 (1.29) | 4.63 (1.26) | 4.77 (1.31)
  Activity Limitation: Day 1 (n=41,41,44,39) | 4.38 (0.83) | 4.07 (0.88) | 4.13 (0.97) | 4.15 (0.91)
  Activity Limitation: Day 29 (n=43,41,44,40) | 4.47 (1.00) | 4.37 (1.07) | 4.42 (1.08) | 4.59 (0.92)
  Activity Limitation: Day 57 (n=44,40,43,45) | 4.57 (1.03) | 4.42 (1.09) | 4.41 (1.14) | 4.74 (0.99)
  Activity Limitation: Day 92 (n=40,42,40,38) | 4.68 (1.19) | 4.89 (1.29) | 4.73 (1.15) | 4.91 (1.04)
  Activity Limitation: Day 127 (n=41,42,44,42) | 4.64 (1.20) | 4.77 (1.32) | 4.62 (1.13) | 4.66 (1.08)
  Activity Limitation: Day 169 (n=41,44,45,44) | 4.68 (1.28) | 4.76 (1.26) | 4.54 (1.31) | 4.70 (1.14)
  Emotional Function: Day 1 (n=41,41,44,39) | 4.30 (1.08) | 4.20 (1.18) | 4.45 (1.10) | 4.29 (1.24)
  Emotional Function: Day 29 (n=43,41,44,40) | 4.64 (1.27) | 4.82 (1.17) | 4.82 (1.22) | 4.88 (1.17)
  Emotional Function: Day 57 (n=44,40,43,45) | 4.85 (1.36) | 4.98 (1.42) | 4.87 (1.24) | 4.99 (1.13)
  Emotional Function: Day 92 (n=40,42,40,38) | 5.00 (1.31) | 5.24 (1.33) | 4.99 (1.45) | 4.98 (1.02)
  Emotional Function: Day 127 (n=41,42,44,42) | 5.08 (1.40) | 5.06 (1.48) | 4.98 (1.40) | 5.28 (1.29)
  Emotional Function: Day 169 (n=41,44,45,44) | 5.05 (1.56) | 5.00 (1.50) | 5.06 (1.39) | 5.13 (1.28)
  Environment stimuli: Day 1 (n=41,41,44,39) | 3.88 (1.28) | 3.55 (1.43) | 3.70 (1.11) | 3.85 (1.10)
  Environment stimuli: Day 29 (n=43,41,44,40) | 4.06 (1.26) | 3.75 (1.48) | 4.13 (1.41) | 4.40 (1.20)
  Environment stimuli: Day 57 (n=44,40,43,45) | 4.07 (1.34) | 4.04 (1.36) | 4.09 (1.43) | 4.37 (1.49)
  Environment stimuli: Day 92 (n=40,42,40,38) | 4.16 (1.56) | 4.44 (1.63) | 4.31 (1.43) | 4.47 (1.47)
  Environment stimuli: Day 127 (n=41,42,44,42) | 4.18 (1.58) | 4.30 (1.57) | 4.15 (1.56) | 4.51 (1.64)
  Environment stimuli: Day 169 (n=41,44,45,44) | 4.13 (1.54) | 4.26 (1.50) | 4.18 (1.76) | 4.45 (1.51)

7. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]) Scores at Day 29, 57, 92, 127 and 169
Description: Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]): a 32-item questionnaire that measures the functional impairments experienced by adult participants including 4 domains (Symptoms, Activity Limitations, Emotional Function, and Environmental Stimuli). Participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score was calculated as the mean response to all questions. The 4 domain scores were the means of the responses to the questions in each of the domains. Overall AQLQ score and 4 domain scores ranged from 7 (no impairment) to 1 (severe impairment). Data collected on Day 1 prior to dosing was considered as baseline
Time Frame: Day 1, 29, 57, 92, 127 and 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
units on a scale
  Overall: Day 29 (n=34,35,37,31) | 0.32 (0.65) | 0.38 (0.64) | 0.39 (0.88) | 0.66 (0.76)
  Overall: Day 57 (n=33,33,35,34) | 0.45 (0.77) | 0.70 (0.99) | 0.38 (0.95) | 0.77 (1.04)
  Overall: Day 92 (n=31,34,35,27) | 0.63 (0.88) | 0.94 (1.21) | 0.52 (1.07) | 1.05 (1.25)
  Overall: Day 127 (n=32,36,34,31) | 0.71 (0.85) | 0.78 (1.21) | 0.49 (1.14) | 1.05 (1.15)
  Overall: Day 169 (n=31,37,37,34) | 0.64 (1.05) | 0.78 (1.19) | 0.56 (1.09) | 0.75 (1.26)
  Symptom: Day 29 (n=34,35,37,31) | 0.31 (0.81) | 0.49 (0.83) | 0.43 (0.83) | 0.62 (0.80)
  Symptom: Day 57 (n=33,33,35,34) | 0.52 (0.86) | 0.87 (1.10) | 0.44 (0.85) | 0.81 (1.11)
  Symptom: Day 92 (n=31,34,35,27) | 0.76 (1.00) | 1.00 (1.32) | 0.61 (1.11) | 1.14 (1.39)
  Symptom: Day 127 (n=32,36,34,31) | 0.85 (1.03) | 0.87 (1.24) | 0.56 (1.14) | 1.24 (1.23)
  Symptom: Day 169 (n=31,37,37,34) | 0.80 (1.06) | 0.86 (1.22) | 0.62 (1.17) | 0.77 (1.34)
  Activity Limitation: Day 29 (n=34,35,37,31) | 0.21 (0.64) | 0.25 (0.69) | 0.32 (0.96) | 0.57 (0.90)
  Activity Limitation: Day 57 (n=33,33,35,34) | 0.28 (0.79) | 0.44 (0.89) | 0.30 (1.08) | 0.71 (1.07)
  Activity Limitation: Day 92 (n=31,34,35,27) | 0.42 (0.81) | 0.80 (1.12) | 0.51 (1.12) | 1.04 (1.26)
  Activity Limitation: Day 127 (n=32,36,34,31) | 0.43 (0.77) | 0.65 (1.20) | 0.45 (1.14) | 0.72 (1.28)
  Activity Limitation: Day 169 (n=31,37,37,34) | 0.38 (1.09) | 0.68 (1.16) | 0.44 (1.09) | 0.65 (1.37)
  Emotional Function: Day 29 (n=34,35,37,31) | 0.50 (0.93) | 0.57 (0.76) | 0.36 (1.04) | 0.86 (0.97)
  Emotional Function: Day 57 (n=33,33,35,34) | 0.69 (1.15) | 0.95 (1.16) | 0.42 (1.15) | 0.86 (1.21)
  Emotional Function: Day 92 (n=31,34,35,27) | 0.87 (1.25) | 1.06 (1.25) | 0.43 (1.26) | 0.93 (1.39)
  Emotional Function: Day 127 (n=32,36,34,31) | 1.02 (1.20) | 0.87 (1.38) | 0.41 (1.32) | 1.32 (1.42)
  Emotional Function: Day 169 (n=31,37,37,34) | 0.88 (1.42) | 0.88 (1.36) | 0.63 (1.20) | 0.95 (1.40)
  Environmental Stimuli: Day 29 (n=34,35,37,31) | 0.40 (0.85) | 0.16 (0.78) | 0.47 (1.18) | 0.76 (0.80)
  Environmental Stimuli: Day 57 (n=33,33,35,34) | 0.36 (0.86) | 0.58 (1.39) | 0.38 (1.27) | 0.65 (1.40)
  Environmental Stimuli: Day 92 (n=31,34,35,27) | 0.54 (0.94) | 0.97 (1.68) | 0.42 (1.17) | 0.94 (1.28)
  Environmental Stimuli: Day 127 (n=32,36,34,31) | 0.64 (1.11) | 0.74 (1.68) | 0.48 (1.45) | 1.02 (1.22)
  Environmental Stimuli: Day 169 (n=31,37,37,34) | 0.52 (1.17) | 0.75 (1.55) | 0.58 (1.30) | 0.74 (1.39)

8. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient Global Impression of Change (PGIC): participant rated instrument to measure participant's change in overall status compared to baseline on a 7-point scale; range from 1 (very much worse) to 7 (very much better).
Time Frame: Day 92 and 169
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
units on a scale
  Day 92 (n=40,42,40,38) | 5.1 (1.1) | 5.3 (1.1) | 5.3 (1.0) | 5.2 (1.2)
  Day 169 (n=42,44,45,44) | 5.1 (1.1) | 5.3 (1.1) | 5.0 (1.0) | 5.1 (1.3)

9. Secondary Outcome: Percentage of Participants With Mean Asthma Control Questionnaire (ACQ) Score Less Than or Equal to 0.75 or ACQ Score Greater Than 0.75 But Less Than 1.5
Description: Percentage of participants with mean Asthma Control Questionnaire (ACQ) score less than or equal to (<=) 0.75 or mean ACQ score greater than (>) 0.75 and less than (<) 1.5 were analyzed. The ACQ is a participant-reported questionnaire to assess the asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Each item was rated on a 7-point Likert scale ranging from 0 (no impairment) to 6 (maximum impairment). Overall ACQ score is the mean of the 6 item scores with a score range of 0 (well controlled) to 6 (extremely poor controlled). Mean ACQ scores of less than or equal to (<=) 0.75 indicated well-controlled asthma, mean ACQ scores greater than (>) 0.75 but less than (<) 1.5 indicated partly controlled asthma.
Time Frame: Day 92 and 169
Population: Evaluable population included all participants who received at least 4 doses of investigational product or received at least 1 dose but discontinued treatment due to safety reasons.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
percentage of participants
  ACQ score<=0.75: Day 92 | 13.0 (19.6) | 19.6 | 11.8 | 17.0
  ACQ score>0.75 and <1.5: Day 92 | 15.2 | 13.0 | 15.7 | 19.1
  ACQ score<=0.75: Day 169 | 13.0 | 19.6 | 13.7 | 19.1
  ACQ score>0.75 and <1.5: Day 169 | 21.7 | 10.9 | 17.6 | 19.1
Statistical Analysis 1: Comparison: Placebo vs CAT-354 150 mg vs CAT-354 300 mg vs CAT-354 600 mg; Test type: Superiority or Other; p = 0.934, Fisher Exact — ACQ score <=0.75, Day 92: Fisher exact test was used to compare all arms
Statistical Analysis 2: Comparison: Placebo vs CAT-354 150 mg vs CAT-354 300 mg vs CAT-354 600 mg; Test type: Superiority or Other; p = 0.592, Fisher Exact — ACQ score <=0.75, Day 169: Fisher exact test was used to compare all arms

10. Secondary Outcome: Serum Concentration for CAT-354
Time Frame: Predose on Day 15, 29, 43, 57, 71 and 85; Day 88, 92, 99, 127, and 169
Population: Pharmacokinetic (PK) population included participants who received CAT-354 and had a sufficient number of serum concentration measurements for computing PK parameters. Here, 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 47 | 51 | 48
microgram per milliliter (mcg/mL)
  Day 15 (n=46,48,48) | 14.5 (5.57) | 27.8 (10.3) | 56.4 (16.0)
  Day 29 (n=45,51,47) | 20.8 (7.20) | 40.2 (15.0) | 81.9 (23.5)
  Day 43 (n=46,50,47) | 26.9 (12.7) | 51.0 (16.0) | 98.5 (33.4)
  Day 57 (n=46,48,46) | 28.4 (11.3) | 58.8 (20.2) | 108 (35.8)
  Day 71 (n=46,49,47) | 29.3 (11.9) | 61.0 (21.4) | 112 (41.2)
  Day 85 (n=45,49,47) | 31.1 (12.5) | 62.0 (23.8) | 120 (44.5)
  Day 88 (n=46,48,45) | 43.4 (15.8) | 85.7 (32.7) | 157 (56.5)
  Day 92 (n=45,46,45) | 42.0 (16.3) | 86.8 (33.1) | 156 (46.6)
  Day 99 (n=46,50,46) | 31.3 (13.0) | 69.3 (27.2) | 125 (41.9)
  Day 127 (n=47,48,47) | 11.5 (6.02) | 22.9 (12.0) | 43.7 (20.5)
  Day 169 (n=47,48,46) | 2.94 (2.23) | 5.87 (3.69) | 10.1 (6.71)

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies to CAT-354 at Any Visit
Time Frame: Day 1, 92 and 169
Population: Safety population included all participants who received any dose of the investigational product. Here, 'N'(number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 47 | 47 | 49 | 47
participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Positive Serum Antibodies to CAT-354 at Any Visit
Time Frame: Day 1, 92 and 169
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 47 | 47 | 49 | 47
percentage of participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and Day 169 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 to 169
Population: Safety population included all participants who received any dose of the investigational product.
Measure: Number; unit: participants
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 47 | 47 | 51 | 48
participants
  TEAEs | 17 | 20 | 25 | 25
  TESAEs | 3 | 2 | 0 | 1

14. Secondary Outcome: Percentage of Participants With at Least 1 Moderate or Severe Exacerbation
Description: Asthma exacerbation was defined as either a progressive increase of asthma symptoms (cough, wheeze, chest tightness, and/or shortness of breath) or a reduction of >= 20 percent (%) in PEF or FEV1 from baseline that did not resolve after the initiation of rescue medications and resulted in an administration of systemic corticosteroids by the investigator or health care provider. Asthma exacerbation severity was classified as: 1) Moderate-worsening symptoms that required systemic corticosteroids. 2) Severe-worsening symptoms that required systemic corticosteroids and hospital admission.
Time Frame: Day 92 and 169
Population: Evaluable population included all participants who received at least 4 doses of investigational product or received at least 1 dose but discontinued treatment due to safety reasons. No separate analyses were performed for moderate and severe exacerbations since only 1 participant had a severe exacerbation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
Percentage of Participants
  Day 92 | 4.3 | 2.2 | 2.0 | 4.3
  Day 169 | 4.3 | 4.3 | 3.9 | 6.4
Statistical Analysis 1: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Day 92: Fisher exact test was used for the analysis
Statistical Analysis 2: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.6022, Fisher Exact — Day 92: Fisher exact test was used for the analysis
Statistical Analysis 3: Comparison: Placebo vs CAT-354 600 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Day 92: Fisher exact test was used for the analysis
Statistical Analysis 4: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Day 169: Fisher exact test was used for the analysis
Statistical Analysis 5: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Day 169: Fisher exact test was used for the analysis
Statistical Analysis 6: Comparison: Placebo vs CAT-354 600 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Day 169: Fisher exact test was used for the analysis

15. Secondary Outcome: Moderate or Severe Asthma Exacerbations Per Person Per Annum
Description: Asthma exacerbation was defined as either a progressive increase of asthma symptoms (cough, wheeze, chest tightness, and/or shortness of breath) or a reduction of >=20% in PEF or FEV1 from baseline that did not resolve after the initiation of rescue medications and resulted in an administration of systemic corticosteroids by the investigator or health care provider. Asthma exacerbation rate, calculated as total asthma exacerbations per person per annum, was assessed based on asthma exacerbation data up to Day 92 and 169 (Rate = mean asthma exacerbations for all participants/X days*365 days, where X = 92 or 169).
Time Frame: Day 1 to Day 92 and Day 169
Population: as for outcome 9
Measure: Mean (Standard Error); unit: asthma exacerbations/person/annum
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
asthma exacerbations/person/annum
  Day 1 to 92 | 0.26 (0.19) | 0.09 (0.09) | 0.08 (0.08) | 0.25 (0.19)
  Day 1 to 169 | 0.23 (0.19) | 0.14 (0.10) | 0.08 (0.06) | 0.19 (0.11)
Statistical Analysis 1: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 0.551, Van Elteren Test — Day 1 to 92: P-value was calculated against placebo group from Van Elteren Test
Statistical Analysis 2: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.492, Van Elteren Test — Day 1 to 92: P-value was calculated against placebo group from Van Elteren Test
Statistical Analysis 3: Comparison: Placebo vs CAT-354 600 mg; Test type: Superiority or Other; p = 0.983, Van Elteren Test — Day 1 to 92: P-value was calculated against placebo group from Van Elteren Test
Statistical Analysis 4: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 0.991, Van Elteren Test — Day 1 to 169: P-value was calculated against placebo group from Van Elteren Test
Statistical Analysis 5: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.900, Van Elteren Test — Day 1 to 169: P-value was calculated against placebo group from Van Elteren Test
Statistical Analysis 6: Comparison: Placebo vs CAT-354 600 mg; Test type: Superiority or Other; p = 0.673, Van Elteren Test — Day 1 to 169: P-value was calculated against placebo group from Van Elteren Test

16. Secondary Outcome: Time to First Moderate or Severe Asthma Exacerbation
Description: Time to first moderate or severe asthma exacerbation was defined as time to first observed progressive increase of asthma symptoms (cough, wheeze, chest tightness, and/or shortness of breath) or a reduction of >=20% in PEF or FEV1 from baseline that did not resolve after the initiation of rescue medications and resulted in an administration of systemic corticosteroids by the investigator or health care provider.
Time Frame: Day 1 to Day 92 and Day 169
Population: as for outcome 9
Measure: Mean (Standard Error); unit: days
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Number analyzed (Participants) | 46 | 46 | 51 | 47
days
  Day 1 to 92 | 89.67 (1.56) | 90.43 (1.32) | 88.16 (2.12) | 89.94 (1.36)
  Day 1 to 169 | 162.24 (3.79) | 163.50 (3.24) | 158.29 (4.41) | 161.21 (3.71)
Statistical Analysis 1: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 0.546, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.534, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.847, Log Rank — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs CAT-354 150 mg; Test type: Superiority or Other; p = 0.987, Log Rank — [p-value comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Placebo vs CAT-354 300 mg; Test type: Superiority or Other; p = 0.992, Log Rank — [p-value comment as in outcome 2, analysis 4]
Statistical Analysis 6: Comparison: Placebo vs CAT-354 600 mg; Test type: Superiority or Other; p = 0.688, Log Rank — [p-value comment as in outcome 2, analysis 4]

ADVERSE EVENTS:
Time Frame: Day 1 to 169
Arm/Group | Placebo | CAT-354 150 mg | CAT-354 300 mg | CAT-354 600 mg
Serious Adverse Events (participants affected / at risk) | 3/47 | 2/47 | 0/51 | 1/48
Other Adverse Events (participants affected / at risk) | 17/47 | 19/47 | 25/51 | 25/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | CAT-354 150 mg (N=47) | CAT-354 300 mg (N=51) | CAT-354 600 mg (N=48)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somatoform disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=47) | CAT-354 150 mg (N=47) | CAT-354 300 mg (N=51) | CAT-354 600 mg (N=48)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (4)
Infusion site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (7) | 0 (0) | 1 (1) | 2 (3)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 2 (3) | 2 (8) | 1 (7)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
H1n1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (5) | 3 (4) | 4 (5)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood chloride increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (3) | 1 (2) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Reticulocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 6 (8) | 1 (1) | 6 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crystalluria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nitrituria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menopausal disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 5 (9) | 5 (6) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (4) | 1 (1) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Labile hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.